CLINICAL TRIAL: NCT04518462
Title: A Phase 3, Randomized, Double Blinded, Active Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of EXPAREL, EXPAREL Admixed With Bupivacaine HCl vs. Bupivacaine HCl Administered as Combined Sciatic (in Popliteal Fossa) and Saphenous (in Adductor Canal) Nerve Blocks for Postsurgical Analgesia in Subjects Undergoing Lower Extremity Surgeries
Brief Title: Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of EXPAREL, EXPAREL Admixed With Bupivacaine HCl vs. Bupivacaine HCl Administered as Combined Sciatic and Saphenous Nerve Blocks for Postsurgical Analgesia in Subjects Undergoing Lower Extremity Surgeries
Acronym: STRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-333
Record Dates: First submitted 2020-08-04; First posted 2020-08-19 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Lower Extremity Surgery; Bunion; Metatarsophalangeal Fushion; Midfoot Fusion; Hindfoot Fushion; Total Ankle Arthroplasty
MeSH Terms: conditions — Bunion | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EXPAREL arm (Experimental): Subjects randomized to this treatment arm will receive 20 mL (266 mg)EXPAREL mixed with 20 mL saline
  Interventions: Drug: Exparel
- EXPAREL admix arm (Experimental): subjects randomized to this treatment arm will receive 20 mL (266 mg)EXPAREL admixed with 20 mL (50 mg) 0.25% bupivacaine HCl.
  Interventions: Drug: Exparel; Drug: Bupivacaine Hydrochloride
- Bupivacaine HCl Arm (Active Comparator): subjects randomized to this treatment arm will receive 40 mL (100 mg)0.25% bupivacaine HCl.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Exparel — EXPAREL (bupivacaine liposome injectable suspension)
  Arms: EXPAREL admix arm; EXPAREL arm
Drug: Bupivacaine Hydrochloride — 0.25% bupivacaine
  Arms: Bupivacaine HCl Arm; EXPAREL admix arm

SUMMARY:
This is a Phase 3, multicenter, randomized, double blinded, active controlled study in approximately 120 subjects undergoing lower extremity surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers ages 18 or older
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
3. Able to provide informed consent, adhere to the study schedule, and complete all study assessments
4. Body Mass Index (BMI) ≥18 and ≤40 kg/m2

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine HCl, nonsteroidal anti-inflammatory drugs [NSAIDs])
2. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post dosing period for pain and which, in the investigator's opinion, may confound the post dosing assessments
3. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
4. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
5. Previous participation in an EXPAREL study
6. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance
7. Currently pregnant, nursing, or planning to become pregnant during the study
8. Clinically significant medical disease that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes diabetic neuropathy, coagulation or bleeding disorders, severe peripheral vascular disease, renal insufficiency, hepatic dysfunction or other conditions that would constitute a contraindication to participation in the study.
9. Currently on a neuromodulating agent neuroleptic agent (e.g., gabapentin, pregabalin [Lyrica], duloxetine [Cymbalta], etc.)
10. Inadequate sensory function on the foot (monofilament test)
11. Chronic opioid use within 30 days prior to randomization (average ≥30 oral morphine equivalents/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - Lotus Clinical Research, Pasadena, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - HD Research, Corp, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL Arm: Subjects randomized to this treatment arm will receive 20 mL (266 mg) EXPAREL mixed with 20 mL saline
  EXPAREL (bupivacaine liposome injectable suspension)
- EXPAREL Admix Arm: subjects randomized to this treatment arm will receive 20 mL (266 mg) EXPAREL admixed with 20 mL (50 mg) 0.25% bupivacaine HCl.
  EXPAREL (bupivacaine liposome injectable suspension)
  Bupivacaine Hydrochloride: 0.25% bupivacaine
- Bupivacaine HCl Arm: subjects randomized to this treatment arm will receive 40 mL (100 mg) 0.25% bupivacaine HCl.
  Bupivacaine Hydrochloride: 0.25% bupivacaine
Period: Overall Study
Arm/Group | EXPAREL Arm | EXPAREL Admix Arm | Bupivacaine HCl Arm
Started | 40 | 41 | 40
Completed | 39 | 40 | 39
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL Arm | EXPAREL Admix Arm | Bupivacaine HCl Arm | Total
Number analyzed (Participants) | 39 | 40 | 40 | 119
Age, Customized [Count of Participants; unit: Participants]
  <45 years | 11 | 14 | 18 | 43
  >/=45 years | 28 | 26 | 22 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 27 | 98
  Male | 4 | 4 | 13 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 15 | 37
  Not Hispanic or Latino | 28 | 26 | 25 | 79
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 11 | 7 | 23
  White | 32 | 26 | 30 | 88
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2
American Society of Anesthesiologists (ASA) Classification [Count of Participants; unit: Participants] — ASA I normal, healthy pt. ASA II mild systemic disease ASA III severe systemic disease ASA IV severe systemic disease that is a constant threat to life
  Participants
    ASA 1 | 15 | 12 | 23 | 50
    ASA 2 | 24 | 26 | 17 | 67
    ASA 3 | 0 | 2 | 0 | 2
    ASA >/= 4 | 0 | 0 | 0 | 0
Height [Number; unit: participants]
  <165 cm | 20 | 21 | 20 | 61
  >/= 165 cm | 19 | 19 | 20 | 58
Weight [Mean (Full Range); unit: kg] | 77.05 [43.5 to 120.2] | 83.03 [49.8 to 117.3] | 77.34 [52.9 to 136.6] | 79.16 [43.5 to 136.6]
Body Mass Index (BMI) kg/m2 [Number; unit: participants]
  <25 kg/m2 | 10 | 9 | 10 | 29
  25- <30kg/m2 | 15 | 10 | 19 | 44
  >/= 30 kg/m2 | 14 | 21 | 11 | 46
Average and worst pain intensity score (NRS) in the last 30 days [Mean (Standard Deviation); unit: score on a scale] — Numerical Rating Scale: an 11 point scale 0=no pain, 10= the worst pain imaginable
  score on a scale
    average NRS | 2.3 (2.53) | 3.2 (2.94) | 2.2 (2.24) | 2.6 (2.60)
    worst NRS | 3.3 (2.64) | 4.5 (3.14) | 3.3 (2.76) | 3.7 (2.88)
Pain Catastrophizing Scale Total Score [Mean (Standard Deviation); unit: score on a scale] — Each question on the Pain Catastrophizing Scale (PCS) is rated from 0 (not at all) to 4 (all the time) total score is from 0-52, with subscale scores assessing rumination, magnification and helplessness.
  score on a scale | 11.7 (11.49) | 13.4 (11.91) | 11.0 (10.68) | 12.0 (11.32)

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of the Analgesic Effect (NRS Pain Intensity) (AUC)
Description: To compare the magnitude of the analgesic effect (NRS pain intensity scores) following a single dose injection of EXPAREL vs. bupivacaine hydrochloride (HCl) when administered as combined sciatic (in the popliteal fossa) and saphenous (in the adductor canal) nerve blocks in subjects undergoing lower extremity surgeries.
  Numerical Rating Scale: an 11 point scale 0=no pain, 10= the worst pain imaginable. The area under the curve (AUC) of the NRS pain intensity scores from 0 to 96 hours post-surgery comparing EXPAREL to 0.25% bupivacaine HCl
Time Frame: Post surgery - 96 hours
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | EXPAREL Arm | EXPAREL Admix Arm | Bupivacaine HCl Arm
Number analyzed (Participants) | 39 | 40 | 40
score on a scale*hours | 298.65 (173.524) | 358.10 (223.610) | 380.05 (220.878)

2. Secondary Outcome: Total Opioid Consumption
Description: Total Opioid Consumption in oral morphine equivalents
Time Frame: 0 hours to 96 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: OMED mg
Arm/Group | EXPAREL Arm | EXPAREL Admix Arm | Bupivacaine HCl Arm
Number analyzed (Participants) | 39 | 40 | 40
OMED mg | 20.68 [13.51 to 31.65] | 23.56 [15.54 to 35.73] | 19.84 [12.72 to 30.96]

3. Secondary Outcome: Time to First Opioid
Description: Time to First Opioid following a single dose of EXPAREL vs. Bupivacain HCl
Time Frame: Post Surgery through Day 14
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | EXPAREL Arm | EXPAREL Admix Arm | Bupivacaine HCl Arm
Number analyzed (Participants) | 39 | 40 | 40
hours | 5.65 [0.72 to 13.55] | 11.93 [5.15 to 16.28] | 16.67 [7.53 to 22.33]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and SAEs were recorded from the time of informed consent through POD 14.
Arm/Group | EXPAREL Arm | EXPAREL Admix Arm | Bupivacaine HCl Arm
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 28/39 | 29/41 | 31/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXPAREL Arm (N=39) | EXPAREL Admix Arm (N=41) | Bupivacaine HCl Arm (N=39)
Constipation (Gastrointestinal disorders) | 9 (9) | 11 (11) | 11 (11)
Nausea (Gastrointestinal disorders) | 8 (11) | 12 (14) | 7 (7)
Vomiting (Gastrointestinal disorders) | 1 (3) | 6 (8) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 10 (10) | 4 (5) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 8 (8) | 9 (9) | 0 (0)
Motor dysfuction (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 5 (8) | 3 (6) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication </= 18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for </=120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT04518462/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT04518462/SAP_001.pdf